CLINICAL TRIAL: NCT05313399
Title: Skeletal and Dentoalveolar Effects of Palatal Crib Versus Bonded Spurs in Early Treatment of Anterior Open Bite Caused by Non-nutritive Sucking Habits: A Randomised Clinical Trial.
Brief Title: Palatal Crib Versus Bonded Spurs in Early Treatment of Anterior Open Bite Caused by Non-nutritive Sucking Habits: RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Reem Hatem Shams (Other)
Responsible Party: Sponsor-Investigator, Reem Hatem Shams, Master Student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 457
Record Dates: First submitted 2022-03-22; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Anterior Open Bite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): the group have open bite caused by non-nutritive sucking habits and treat them with palatal crib.
  Interventions: Device: Palatal Crib
- experimental group (Experimental): the group have open bite caused by by non-nutritive sucking habit and treat them with bonded spur.
  Interventions: Device: bonded spur

INTERVENTIONS:
Device: Palatal Crib — An intraoral appliance approach can be used as an adjunct method to stop the habit. Appliances consisting of cribs in the anterior region are very efficient as reminders and physical restrainers. The palatal crib works as an obstacle in non-nutritive sucking and maintains the tongue in a more retruded position, halting its interposition between the incisors.
  Arms: control group
Device: bonded spur — Spur appliances change tongue action, close the open bite, and boost treatment stability, as it induces a permanent modification of the tongue's anterior rest posture by altering orofacial function, resulting in a change in form. Finally, the spur adjusts the sensory input to the brain. This proprioceptive change leads to an altered motor response, resulting in a new normal tongue rest posture (change in function) that allows the incisors to erupt
  Arms: experimental group

SUMMARY:
The study evaluates the effects of palatal crib versus bonded spurs in the early treatment of anterior open bite caused by non-nutritive sucking habits.

DETAILED DESCRIPTION:
Habit is an unintentionally performed repeated activity. Development of habit is considered a part of the natural progression of maturation in children between infancy and three years of age, after this period, it is assumed to be unnatural. The most familiar and earliest noted habit is thumb sucking. It develops during infancy as a rooting reflex, after it ceases around three years of age .

Thumb sucking is defined as the placement of the thumb or one or more fingers in different depths into the mouth ). It emerges in two forms: nutritive and non-nutritive, where the first gives nourishment and the second implements a sense of security and amenity. It is common in children and is reported to be harmless for up to five years of age .

There is an association between the habit of thumb sucking and the development of skeletal open-bite among children. Anterior open bites (AOBs) are defined as an occlusion in which the lower incisors are not overlapped in the vertical plane by the upper incisors and do not occlude with them when the posterior teeth are in maximum intercuspation . Anterior open bite due to thumb sucking, and a secondary tongue thrust exaggerates the condition . If identified early, this can be avoided and appropriate treatment is delivered.

Approaches for habit intervention include counseling, positive reinforcement, a calendar with rewards, an adhesive bandage, bitter nail polish, long sleeves, and appliance therapy. It is recommended to start with the least invasive methods before using habit-breaking appliances. Habit-breaking appliances are either fixed or removable. Fixed appliance therapy may be considered after the age of 4 years. Appliances consisting of cribs in the anterior region are very efficient as reminders and physical restrainers . The palatal crib works as an obstacle in non-nutritive sucking and maintains the tongue in a more retruded position, halting its interposition between the incisors. Spur appliances change tongue action, close the open bite, and boost treatment stability, as it induces a permanent modification of the tongue's anterior rest posture by altering orofacial function, resulting in a change in form. Finally, the spur adjusts the sensory input to the brain. This proprioceptive change leads to an altered motor response, resulting in a new normal tongue rest posture (change in function) that allows the incisors to erupt.

ELIGIBILITY:
Inclusion Criteria:

1. Children with nonnutritive sucking habits and/or tongue thrusting from 6 years to 11 years old.
2. Angle Class I malocclusions.
3. Anterior open bite equal to or greater than 1 mm.
4. Maxillary and mandibular permanent central incisors fully erupted (children in the first transitional period were eligible for treatment when the maxillary lateral incisors were beginning to erupt, and the maxillary central incisors were still showing an open bite).

Exclusion Criteria:

1. Children with loss of permanent teeth.
2. Crowding, maxillary constriction, or posterior crossbites.
3. Previous orthodontic treatment.
4. Presence of craniofacial anomalies or syndromes.
5. Tooth agenesis.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Overbite distance correction in millimeter | 12 months
  Digital dental model will be scanned using medit software to detect the changes that occur in the vertical distance ( in millimeter ) between incisal edges of the most erupted maxillary and mandibular central incisors in relation to the occlusal plane.

SECONDARY OUTCOMES:
Changes in maxillary mandibular plane angle | 12 months
  standardised lateral cephalometric radiographs will be taken, and the variables will be digitally traced using Dolphin Imaging Software Version 11.5
Patient acceptance | 1 month
  1. The questionnaire is consisted of 5 questions and has space for additional patient comments.
  2. The variables in the first four questions will assess speaking, eating, esthetics, and pain.
  3. The rating scale that will be used to quantify the effect of the spurs and the palatal crib on these variables 1 (easy), 2 (neutral), and 3 (difficult).
  4. The 5th question on the survey will assess the time needed by the patients to adjust the presence of the two appliances. Possible answers are 2 days or less, 1 week, 2 weeks, and longer.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Elkhadem, Ass. professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leite JS, Matiussi LB, Salem AC, Provenzano MG, Ramos AL. Effects of palatal crib and bonded spurs in early treatment of anterior open bite: A prospective randomized clinical study. Angle Orthod. 2016 Sep;86(5):734-9. doi: 10.2319/031815-170.1. Epub 2015 Dec 31. PMID 26719946
- See also: correction of open bite caused by non-nutritive sucking habit by using palatal crib and bonded spur — https://pubmed.ncbi.nlm.nih.gov/PMC8600830/